CLINICAL TRIAL: NCT05391074
Title: Pilot Study to Evaluate the Safety and Efficacy of Oral Therapy With Postbiotics in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration, Myopia, or Angioid Streaks
Brief Title: Oral Postbiotics in Patients With Macular Atrophy
Acronym: REVERS-GA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de la Macula y la Retina (Other)
Collaborators: Igen BioLab SLU (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InstitutMaculaRetina
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
Keywords: postbiotics; microbiota; microbiome; geographic atrophy; atrophic AMD; AMD; age-related macular degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with GA secondary to AMD, myopia or angioid streaks (Experimental): postbiotics (IGENH35.3A) with vitamins (AREDS formulation and recommended daily dose)
  Interventions: Dietary Supplement: postbiotics (IGENH35.3A); Dietary Supplement: vitamins (AREDS formulation and recommended daily dose)

INTERVENTIONS:
Dietary Supplement: postbiotics (IGENH35.3A) — postbiotics to induce microbiota epigenetic factors
Dietary Supplement: vitamins (AREDS formulation and recommended daily dose) — vitamins (AREDS to prevent AMD progression

SUMMARY:
A pilot study to evaluate the safety and efficacy of oral therapy with Postbiotics in patients with geographic atrophy secondary to age-related macular degeneration, myopia, or angioid streaks.

DETAILED DESCRIPTION:
A pilot study to evaluate the safety and efficacy of oral therapy with Postbiotics in patients with geographic atrophy (GA) secondary to age-related macular degeneration, myopia or angioid streaks.

The study's main objective is to evaluate if oral postbiotic therapy will induce epigenetic factors that would impact the progression of the GA, and it will compare the rate of growth of GA from the Baseline to 12 months, to the rate shown during the 12 months before Baseline.

ELIGIBILITY:
Inclusion Criteria:

* patients with GA secondary to AMD, myopia or angioid streaks
* with 12 months of previous follow-up,
* and a known progression of >0,20mm/year as per SQRT

Exclusion Criteria:

- history of choroidal neovascularization in the study eye

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
rate of growth of geographic atrophy (GA) as per SQRT (square roor transformation) of area of GA measured in FAF, (fundus autofluorescence) | 12 months
  rate of growth of GA as per SQRT of FAF area compared to rate of growth of the previous year
safety and tolerability | 12 months
  safety and tolerability of daily dosing of oral postbiotics assessed by number of patients with clinically significant changes of a combination of ocular and/or non-ocular adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Monés, MD, PhD, Principal Investigator — Institut de la Màcula
Locations (1):
- Institut de la Màcula, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No